CLINICAL TRIAL: NCT00339716
Title: Scientific Protocol for the Study of Thyroid Cancer and Other Thyroid Disease in Belarus Following the Chernobyl Accident
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999995021; OH95-C-N021
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Thyroid Cancer; Non-Cancer Thyroid Disease; Non Thyroid Cancer
Keywords: Cohort; Radiation; In Utero
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Belarus in utero: subjects exposed to I131 in utero
- Main BelAm: subjects exposed to I131 at age less than 18 year

SUMMARY:
Iodine-131(131I) and other radioisotopes of Iodine are contained in fallout from atmospheric nuclear weapons tests and are among the radionuclides most likely to be released in a nuclear reactor accident. In spite of nearly 50 years of experience, the risk of thyroid disease, especially thyroid cancer, attributable to exposure to 131I remains unknown, although the carcinogenic potential of x-ray and gamma-ray exposure of the thyroid is reasonably well known. The available data also indicate that children face greater risks of radiation-induced thyroid cancer than do adults.

The nuclear power plant accident at Chernobyl released large quantities of 131I and other radioisotopes of iodine into the atmosphere, contaminating thousands of square kilometers and exposing millions of people. It is proposed that a well-defined subset of Belarussian children aged 0-18 years at the time of the accident be examined by well-trained specialists for thyroid disease at least biennially for up to 30 years. A cohort of 15,000 children has been identified, all of whom had their thyroids measured for radioactivity during the weeks immediately following the accident. Under a rigid research protocol these children will receive complete diagnostic thyroid examinations, including palpation, ultrasound scanning, thyroid hormone and other laboratory tests, and fine-needle aspiration, as appropriate. Cancer will be determined by expert pathology examination of tissue. In addition to the analysis of thyroid radiation measurements made in May-June, 1986, efforts will be made to reconstruct each person's exposure and to estimate the radiation doses to the thyroid. This will involve the reconstruction of deposition patterns and environmental pathways of the radioiodines, and of the location, dietary characteristics, and lifestyle of each person throughout the exposure period.

The data will be analyzed to evaluate the relationship, if any, between thyroid disease, especially cancer, and the radiation dose to the thyroid, with emphasis on the dose from 131I. The primary focus will be on dose-response analyses of person-year incidence data with stratification by sex, age at exposure, geographic area, time, and age at risk. Confounding factors, e.g., use of potassium iodide (KI) as a prophylactic measure, will be evaluated and controlled in the analysis, and the uncertainty of the dose estimates will be taken into account.

In addition to producing risk coefficients for thyroid cancer and other thyroid diseases in children as a function of sex and age at the time of exposure, it is expected that the analyses will contribute new knowledge of the carcinogenic effectiveness of 131I in comparison with that of x-ray and gamma radiation. This information will fill a major gap in the world's knowledge of radiation effects, and will provide guidance for radiation protection and public health policies wherever nuclear reactors are in operation.

DETAILED DESCRIPTION:
The nuclear power plant accident at Chornobyl released large quantities of Iodine-131 and other radioisotopes of iodine into the atmosphere, contaminating thousands of square kilometers and exposing millions of people. For this study, a well-defined subset of Belarusian children under age 18 years at the time of the accident were identified and examined by well-trained specialists for thyroid disease every two years for three cycles. The study is a collaborative effort of researchers in Belarus and the United States.

<TAB>

The cohort includes approximately 12,000 persons who were children in 1986, all of whom had their thyroids measured for radioactivity during the weeks immediately following the accident. Under a rigid research protocol these subjects received diagnostic thyroid examinations, including palpation, ultrasound scanning, thyroid hormone and other laboratory tests. If indicated, they were referred for a fine-needle aspiration biopsy. Interview information regarding residential, health, diet and lifestyle history are also collected. All subjects were followed for thyroid cancer morbidity and mortality. Overall, 163 cancers were identified. Interviews with mothers of the subjects who were less than 10 years of age at the time of the accident whose memory of events proved inadequate increased the total accrual to 13,552.

Based on thyroid radiation measurements made in May-June, 1986, and other information (reconstruction of deposition patterns and environmental pathways of the radioiodines, and of the location, dietary characteristics, and lifestyle of each person throughout the exposure period), each person s radiation dose to the thyroid was estimated.

The aim of the study is to assess the early and late morphologic and functional changes in the thyroid glands of young persons exposed to radiation from radioactive materials released as a consequence of the Chornobyl nuclear power plant accident, with emphasis on dose- and time-specific changes.

Active screening for thyroid cancers ended in September 2006. The third and final thyroid screening examinations were completed in September 2006, identifying 163 cases of thyroid cancer during the examination period. Subject accrual through screening is no longer ongoing. Thyroid and other cancer case ascertainment is underway by linkage to the Belarusian Cancer Registry. A paper has been published on the radiation dose response for prevalent thyroid cancer and analyses of incident cancer cases and other thyroid disease are ongoing.

ELIGIBILITY:
* INCLUSION CRITERIA:

We will include about 3,000 individuals born in Belarus from April, 26, 1986 through March, 31, 1987 who were exposed to internal and external sources of ionizing radiation during prenatal and early postnatal periods due to the Chernobyl fallout.

EXCLUSION CRITERIA:

For the purpose of individual dose reconstruction we need to establish child-mother pair for each cohort member and conduct personal dosimetric interview with child s mother. We anticipate that some of the eligible subjects will be deceased at the time of the cohort construction. Deceased subjects will not be included in the cohort. Excluded from the interview study and the subsequent follow-up study will be those who are deceased, cannot be located, refuse to participate in the study, or do not provide informed consent.

Ages: 30 Years to 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects exposed to I131 at age less than 18 years, and subjects exposed to I131 in utero
Sampling Method: Non-Probability Sample
Enrollment: 19456 (Actual)
Dates: Start 1994-03-21 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Radiation-related risk of benign and malignant thyroid disease | 2-3 years after initiation of study
  radiation risk estimate

CONTACTS AND LOCATIONS:
Overall Officials: Kiyohiko Mabuchi, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- Belarus (2):
  - Republican Resear ch Center for Radiation Medicine and Human Ecology, Homyel
  - Ministry of Health Republic of Belarus, Minsk

REFERENCES:
- [Background] Drozdovitch V, Minenko V, Golovanov I, Khrutchinsky A, Kukhta T, Kutsen S, Luckyanov N, Ostroumova E, Trofimik S, Voilleque P, Simon SL, Bouville A. Thyroid Dose Estimates for a Cohort of Belarusian Children Exposed to (131)I from the Chernobyl Accident: Assessment of Uncertainties. Radiat Res. 2015 Aug;184(2):203-18. doi: 10.1667/rr13791.1. Epub 2015 Jul 24. PMID 26207684
- [Background] Zablotska LB, Nadyrov EA, Polyanskaya ON, McConnell RJ, O'Kane P, Lubin J, Hatch M, Little MP, Brenner AV, Veyalkin IV, Yauseyenka VV, Bouville A, Drozdovitch VV, Minenko VF, Demidchik YE, Mabuchi K, Rozhko AV. Risk of thyroid follicular adenoma among children and adolescents in Belarus exposed to iodine-131 after the Chornobyl accident. Am J Epidemiol. 2015 Nov 1;182(9):781-90. doi: 10.1093/aje/kwv127. Epub 2015 Oct 5. PMID 26443421
- [Background] Little MP, Kwon D, Zablotska LB, Brenner AV, Cahoon EK, Rozhko AV, Polyanskaya ON, Minenko VF, Golovanov I, Bouville A, Drozdovitch V. Impact of Uncertainties in Exposure Assessment on Thyroid Cancer Risk among Persons in Belarus Exposed as Children or Adolescents Due to the Chernobyl Accident. PLoS One. 2015 Oct 14;10(10):e0139826. doi: 10.1371/journal.pone.0139826. eCollection 2015. PMID 26465339